CLINICAL TRIAL: NCT04714203
Title: Assessment of the Prevalence of Sarcopenia in Early Palliative Cancer Patients
Acronym: SPACE
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Responsible Party: Sponsor
Other Study IDs: WP-2019-04
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort: Sarcopenia assessment
  Interventions: Other: sarcopenia assessment

INTERVENTIONS:
Other: sarcopenia assessment — evaluation of sarcopenia status

SUMMARY:
Cancer is one of the leading causes of death in the world after cardiovascular disease (8.7 million deaths in 2015 for 17.5 million cases) 1. Despite a great deal of progress in disease detection and treatment, the incidence of cancer is steadily increasing (+ 33% in 2015) and particularly in certain locations (pancreas, lungs, brain and stomach), including risk factors are not always identified.

Advanced stage cancer (= metastatic) is most often incurable with the exception of germ cell tumors. Palliative care is then most often offered. Palliative care favors the patient's quality of life as a whole (medical, physical, psychological and social).

The symptoms most often reported by patients are: pain, fatigue, decreased appetite, nausea, and are directly related to phenomena such as cachexia, loss of autonomy and deterioration of psychological state, resulting in decreased overall survival. Chemotherapies and targeted therapies (immunotherapy, hormonal therapy, participation in a clinical trial) can provide a benefit in quality of life and survival only in the early phase (little benefit in the terminal phase).

Other prognostic factors can impact the quality of life and overall survival in these situations: sarcopenia and disorders of nutritional status (obesity, undernutrition).

The study of sarcopenia by CT scan of patients in a palliative situation is still too scarce. Sarcopenia is an often underestimated event and is associated with older age, co-morbidities, increased infectious complications, and early mortality.

The study of the prevalence of sarcopenia by CT scan would confirm its prognostic impact in a palliative situation.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years old,
* patient with solid cancer diagnosed with metastatic disease,
* having had a biological assessment and a CT scan in the month preceding the medical consultation,
* and whose prognosis is considered palliative

Exclusion Criteria:

* age <18 years old,
* adults under guardianship measure,
* pregnancy or breastfeeding in progress,
* malignant hemopathies,
* metastatic germ cell tumors,
* non-metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include all patients diagnosed with metastatic disease (either present at diagnosis or occurring after an initially localized cancer).
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of sarcopenia | 1 month
  Number of patients with sarcopenia in the numerator out of the total number of patients included in the study in the denominator

SECONDARY OUTCOMES:
Prevalence of undernutrition | 1 month
  Number of patients with nutritional disorders at inclusion in numerator out of the number of patients followed in denominator
Overall survival | 6 months
  Time between the inclusion date and the date of death regardless of the cause or the date of the latest news if the patient is censored
Progression free survival | 6 months
  Time between the inclusion date and the date of the first examination showing Time disease progression or the date of death if the patient is deceased or the date of the latest news if the patient is censored
Event free survival | 6 months
  Time between the date of inclusion and the date of the first event identified or the date of death if the patient is deceased or the date of the latest news if the patient is censored
Correlation between PRONOPALL score and sarcopenia | 1 months
  Calculation of PRONOPALL score (high score corresponds to a worse situation)

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DU, MD, Principal Investigator — Clinique Victor Hugo/Centre Jean Bernard
Locations (1):
- Clinique Victor Hugo / Centre Jean Bernard, Le Mans, France

IPD SHARING:
Plan to Share IPD: No